CLINICAL TRIAL: NCT03361826
Title: Magnetic Seizure Therapy for the Treatment of Treatment-Resistant Depression and Suicidal Ideation in Borderline Personality Disorder
Brief Title: Magnetic Seizure Therapy for the Treatment of Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Daniel Blumberger, Chair, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 053/2015
Record Dates: First submitted 2017-10-31; First posted 2017-12-05 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Borderline Personality Disorder
Keywords: Magnetic seizure therapy (MST); Treatment resistance; Open-label trial; Borderline Personality Disorder; Suicidal Ideation; Treatment-resistant depression; Dialectical behavior therapy (DBT); MST + DBT; Neuroimaging-based biomarkers
MeSH Terms: conditions — Borderline Personality Disorder; Suicidal Ideation; Depressive Disorder, Treatment-Resistant; Myeloproliferative Syndrome, Transient; Maple syrup urine disease, type 2 | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Using a case-control design, the investigators will compare individuals receiving MST and DBT with matched patient control group receiving DBT alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DBT Only (Other): Dialectical behavior therapy (DBT) is a specific type of cognitive-behavioral psychotherapy developed to help better treat borderline personality disorder.
  Interventions: Behavioral: DBT
- MagPro MST with Cool TwinCoil + DBT (Experimental): MST treatments will be administered using the MagPro MST with Cool TwinCoil. Moderate-to-highly suicidal patients with BPD beginning dialectical behavioural therapy (DBT) will be recruited using a case-control design, comparing individuals receiving MST and DBT with matched patient control group receiving DBT alone.
  Interventions: Device: MagPro MST with Cool TwinCoil; Behavioral: DBT

INTERVENTIONS:
Device: MagPro MST with Cool TwinCoil — MST treatments will be administered using the MagPro MST with Cool TwinCoil. The investigators will evaluate the effectiveness of MST for reducing suicidality and depressive symptoms in an open-label clinical trial of up to 15 treatment sessions. Moderate-to-highly suicidal patients with BPD beginning dialectical behavioural therapy (DBT) will be recruited using a case-control design, comparing individuals receiving MST and DBT with matched patient control group receiving DBT alone.
  Other Names: Magnetic Seizure Therapy (MST)
  Arms: MagPro MST with Cool TwinCoil + DBT
Behavioral: DBT — Dialectical behavior therapy (DBT) is a specific type of cognitive-behavioral psychotherapy developed to help better treat borderline personality disorder. Moderate-to-highly suicidal patients with BPD beginning dialectical behavioural therapy (DBT) will be recruited using a case-control design, comparing individuals receiving MST and DBT with matched patient control group receiving DBT alone.
  Other Names: Dialectical behavior therapy (DBT)

SUMMARY:
Suicide is a major public health crisis for which effective new interventions are needed. An innovative new brain stimulation technique called magnetic seizure therapy (MST) shows promise for treating suicidal thinking in chronically depressed individuals. Using a high-risk cohort of suicidal patients with borderline personality disorder (BPD) and treatment resistant major depressive disorder (MDD), this study will evaluate the effectiveness of MST for reducing suicidality and depressive symptoms in an open-label clinical trial of up to 15 treatment sessions. Based on research showing that functioning of the dorsolateral prefrontal cortex (DLPFC) may be disrupted in BPD and place individuals at risk for suicide, the DLPFC will be targeted for stimulation. Moderate-to-highly suicidal patients with BPD beginning dialectical behavioural therapy (DBT) will be recruited using a case-control design, comparing individuals receiving MST and DBT with matched patient control group receiving DBT alone.

DETAILED DESCRIPTION:
MST is a novel modification of electroconvulsive therapy (ECT) with the potential for similar clinical effectiveness, fewer side-effects and a more rapid return of orientation and shorter duration of post-ictal confusion. In the proposed study, the investigators will evaluate the clinical effectiveness of MST for the treatment of treatment-resistant depression (TRD) and suicidal ideation in patients with BPD. The study will use a case-control design comparing symptom reports (depression severity and suicidal ideation) and cognitive functioning between outpatients receiving MST plus dialectical behavioral therapy (DBT) and matched patient controls receiving DBT alone. To evaluate potential biomarkers that may underlie the anticipated clinical benefits of MST, functional magnetic resonance imaging (fMRI) will be used to measure activation of the DLPFC and associated neural circuits subserving emotion regulation and cognitive functioning (e.g., impulse control, episodic memory) in BPD.

Objective 1: To evaluate the efficacy of MST as a treatment for suicidal ideation and TRD in BPD.

Hypothesis 1: MST will demonstrate substantial efficacy on objective measures of suicidal ideation and depression.

Objective 2: To evaluate the effects of MST on cognitive functioning in patients with BPD.

Hypothesis 2: MST will have limited, if any, effects on performance on standard neuropsychological measures of attention, memory and executive functioning in patients with BPD.

Objective 3: To explore potential neuroimaging-based biomarkers that may index any changes in suicidal ideation and depression that result from treatment with MST.

Hypothesis 3: On neuroimaging tasks assessing emotion processing and cognitive functioning, patients receiving DBT+MST will show increased activity in bilateral DLPFC after treatment relative to pre-treatment baseline activation, and more activation in this region than patients in DBT without concurrent MST (DBT-only).

ELIGIBILITY:
Inclusion Criteria:

* MST+DBT Group

  1. English-speaking and able to provide informed consent to participate in the study
  2. Female and between the ages 18 and 50 years
  3. Current DSM-IV (Diagnostic and statistical manual of mental disorders-IV) diagnosis of BPD based on the International Personality Disorder Examination BPD Section (IPDE-BPD)
  4. Current DSM-IV diagnosis of a non-psychotic, major depressive episode, as part of a broader diagnosis of MDD (single episode or recurrent episode), based on the Structured Clinical Interview for DSM-IV Axis I Disorders-Patient Edition (SCID-I/P)
  5. Score > 9 (equivalent to moderate-to-severe suicidal ideation) on the Modified Suicidal ideation Scale for at least the two weeks prior to enrolling in the study
  6. Hamilton Rating Scale for Depression (HRSD-24) score > 22 (classified as Very Severe Depression)
  7. Failed to achieve a clinical response to adequate treatment trials of two or more antidepressants during the current depressive episode OR have been unable to tolerate at least two antidepressants as assessed by the Antidepressant Treatment History Form (ATHF)
  8. Deemed appropriate to receive ECT as assessed by an ECT attending psychiatrist and an anesthesiologist
  9. Meets the MST safety criteria
  10. Agreeable to keeping their current antidepressant treatment (if any) constant during the intervention (unless clinically indicated)
  11. Has a close family member, friend, partner, or qualified chaperone able and willing to accompany the patient home after each MST treatment session and
  12. Able to adhere to the intervention schedule.
* DBT-Only Group

  1. English-speaking and able to provide informed consent to participate in the study
  2. Female and between the ages 18 and 50 years
  3. Current DSM-IV diagnosis of BPD based on the International Personality Disorder Examination BPD Section (IPDE-BPD)
  4. Current DSM-5 diagnosis of a non-psychotic, major depressive episode, as part of a broader diagnosis of MDD (single episode or recurrent episode), based on the Structured Clinical Interview for DSM-IV Axis I Disorders--Patient Edition (SCID-I)
  5. Score > 9 (equivalent to moderate-to-severe suicidal ideation) on the Modified Suicidal ideation Scale for at least the two weeks prior to enrolling in the study
  6. Baseline Hamilton Rating Scale for Depression (HRSD-24) score > 22
  7. Failed to achieve a clinical response to adequate treatment trials of two or more antidepressants during the current depressive episode OR have been unable to tolerate at least two antidepressants as assessed by the Antidepressant Treatment History Form (ATHF)
  8. Agreeable to keeping their current antidepressant treatment (if any) constant during the study (unless clinically indicated)

Exclusion Criteria:

* MST+DBT Group

  1. Acute suicidal intent that requires hospitalization to protect harm to self
  2. Any unstable medical and/or neurological condition
  3. Currently pregnant or lactating, or intention to get pregnant during the duration of the study
  4. Not considered sufficiently physically healthy to undergo general anesthesia for any reason
  5. Any significant neurological disorder or condition likely to be associated with increased intracranial pressure or cognitive impairment (e.g., a space occupying brain lesion, a history of stroke, a cerebral aneurysm, a seizure disorder, Parkinson's disease, Huntington's chorea, multiple sclerosis)
  6. Medical condition, medication, or laboratory abnormality that could cause a major depressive episode or significant cognitive impairment in the opinion of the investigator (e.g., hypothyroidism with low thyroid-stimulating hormone (TSH), rheumatoid arthritis requiring high dose prednisone, or Cushing's disease)
  7. Current diagnosis of delirium, dementia or another cognitive disorder secondary to a general medical condition
  8. Diagnosis of a developmental disorder (e.g. Down syndrome, autism-spectrum disorder)
  9. Non-correctable clinically significant sensory impairment (i.e., cannot hear or see well enough to complete the neuropsychological tests)
  10. Lower than eighth-grade reading level as assessed by the Wide Range Achievement Test-Fourth Edition
  11. Alcohol or substance use disorder (relating to opioids or cocaine) currently or within the past 1 month
  12. Diagnosis of a DSM-5 psychotic disorder
  13. Demonstrated a lack of response to ECT during the current or prior depressive episode.
  14. Requires a benzodiazepine with a dose equivalent to lorazepam 2 mg/day or higher or any anticonvulsant due to the potential of these medications to limit the efficacy of both MST and ECT
  15. Intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
  16. Has sustained a moderate-to-severe head injury (defined as ≥ 20 min loss of consciousness and/or > 24 hrs post-traumatic amnesia); or
  17. Does not qualify for MRI scanning
* DBT-Only Group

  1. Acute suicidal intent that requires hospitalization to protect harm to self
  2. Any unstable medical and/or neurological condition
  3. Currently pregnant or lactating, or intention to get pregnant during the duration of the study
  4. Any significant neurological disorder or condition likely to be associated with increased intracranial pressure or cognitive impairment (e.g., a space occupying brain lesion, a history of stroke, a cerebral aneurysm, a seizure disorder, Parkinson's disease, Huntington's chorea, multiple sclerosis)
  5. Medical condition, medication, or laboratory abnormality that could cause a major depressive episode or significant cognitive impairment in the opinion of the investigator (e.g., hypothyroidism with low TSH, rheumatoid arthritis requiring high dose prednisone, or Cushing's disease)
  6. Current diagnosis of delirium, dementia or another cognitive disorder secondary to a general medical condition
  7. Diagnosis of a developmental disorder (e.g. Down syndrome, autism-spectrum disorder)
  8. Non-correctable clinically significant sensory impairment (i.e., cannot hear or see well enough to complete the neuropsychological tests)
  9. Lower than eighth-grade reading level as assessed by the Wide Range Achievement Test--Fourth Edition
  10. Alcohol or substance use disorder (relating to opioids or cocaine use) currently or within the past 1 month
  11. Diagnosis of a DSM-5 psychotic disorder
  12. Intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
  13. Has sustained a moderate-to-severe head injury (defined as ≥ 20 min loss of consciousness and/or > 24 hrs post-traumatic amnesia)
  14. Does not qualify for MRI scanning

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 27 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Improvement in symptom severity of depression as measured by the Hamilton Rating Scale for Depression - 24 | 5 weeks
  Hamilton Rating Scale for Depression (24-item version)
  * This scale is used to quantify the severity of symptoms of depression
  * Scale range: 0-76 (total score)
  * Lower scores indicate lower severity of depressive symptoms (i.e., better outcome)
  * Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)
Improvement in symptom severity of Suicidal Ideation as measured by the Modified Scale for Suicidal Ideation | 5 weeks
  Modified Scale for Suicidal Ideation
  * This scale is used to assess the presence or absence of suicidal ideation and the degree of severity of suicidal ideas
  * Scale range: 0-54 (total score)
  * Lower scores indicate lower severity of suicidal ideation (i.e., better outcome)
  * Higher scores indicate higher severity of suicidal ideation (i.e., worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Blumberger, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital — http://www.camh.net/research